CLINICAL TRIAL: NCT00742352
Title: PET FDG Assessment of Change in Atherosclerotic Plaques After Chemotherapy
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Tel-Aviv Sourasky Medical Center (Other Government)
Responsible Party: Prof. Einat Even-Sapir, Tel-Aviv Sourasky Medical Center
Other Study IDs: TASMC-08-EES-253-CTIL
Record Dates: First submitted 2008-08-25; First posted 2008-08-27 (Estimated); Last update posted 2008-09-09 (Estimated); Status verified 2008-08

CONDITIONS: Atherosclerosis
MeSH Terms: conditions — Atherosclerosis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (2):
- Breast cancer patients
- Lung cancer patients

SUMMARY:
The purpose of this study is to determine whether chemotherapy induces regression in atherosclerotic plaques in oncologic patients already undergoing PET FDG as part of their routine assessment.We will use PET FDG to assess whether the inflammation in atherosclerotic plaques is affected by chemotherapy and anti angiogenic therapy.

ELIGIBILITY:
Inclusion Criteria:

* Women over the age of 65 diagnosed with metastatic breast cancer
* Men over the age of 65 diagnosed with lung cancer

Exclusion Criteria:

* Patients under the age of 65
* Patients diagnosed with chronic inflammatory disease or chronic infection
* Patients taking steroids and NSAIDS on a regular basis

Min Age: 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Study Population: Breast cancer patients at the Tel-Aviv Sourasky Medical Center Lung cancer patients at the Tel-Aviv Sourasky Medical Center
Sampling Method: Non-Probability Sample
Enrollment: 40 (Estimated)
Dates: Start 2008-09

CONTACTS AND LOCATIONS:
Locations (1):
- Tel-Aviv Sourasky Medical Center, Tel Aviv, Israel